CLINICAL TRIAL: NCT04513600
Title: Transthyretin Amyloid Cardiomyopathy: Stabilization Assessed by Cardiac Magnetic Resonance
Brief Title: ATTR-Cardiomyopathy Stabilization Following Tafamidis Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christ Hospital (Other)
Collaborators: The Cleveland Clinic (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Dr. Wojciech Mazur, Director of Advanced Cardiac Imaging, The Christ Hospital
Other Study IDs: 20-02
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Lab work: Hs- Troponin, Serum N-terminal-proBNP CMR: Native T1, Native T2, extracellular volume, strain and strain rate.
  Other Names: Blood sample

SUMMARY:
The study will investigate the stabilization effects of Tafamidis utilizing cardiac imaging cardiac magnetic resonance imaging (CMR). The investigators propose to pursue the following specific aims:

1. Utilize cardiac magnetic resonance to assess stabilization of ATTR after Tafamidis therapy based on extracellular volume mapping.
2. Investigate left ventricular myocardial mass, native T1, T2, and extracellular volume mapping after 12 month follow-up.
3. Utilize cardiac magnetic resonance feature tracking at baseline and at 12 month follow-up.

DETAILED DESCRIPTION:
The investigators hypothesize that participants with earlier stages (NYHA Class I and Class II) of ATTR wild type and ATTR mutant will demonstrate stabilization of ATTR following 1 year of Tafamidis.

The investigators propose to pursue the following specific aims:

1. Utilize cardiac magnetic resonance to assess stabilization of ATTR after Tafamidis therapy based on extracellular volume mapping.
2. Investigate left ventricular myocardial mass, native T1, T2, and extracellular volume mapping after 12 month follow-up.
3. Utilize cardiac magnetic resonance feature tracking at baseline and at 12 month follow-up.

The investigators will enroll 131 participants with confirmed ATTR. Participants will be screened to exclude light chain amyloidosis by either measuring the proportion of kappa: lambda light chains with the serum free light chain assay, and tested for immunofixation electrophoresis of serum and urine. Once participants has confirmed diagnosis of ATTR (pyrophosphate scan positive scoring >1.5 ratio) and undergone baseline testing participants will be ask to enroll in the study. Genetic testing will performed to further distinguish between mutation and wild type. All participants will be required to sign informed consent agreeing to follow up testing at 1 year.

Participants will undergo a baseline cardiac magnetic resonance imaging for the purpose of evaluating native T1, T2, first pass perfusion, and extracellular volumes for patients with glomerular filtration rate >30. Patients with glomerular filtration rate <30 will only have native T1 and T2 values evaluated. If participants undergo implanted cardiac device during Tafamidis therapy, follow up cardiac magnetic resonance imaging will only evaluate featuring tracking and left ventricular mass. Left ventricular mass and cardiac magnetic feature tracking values will be extracted from all cardiac magnetic resonance imaging studies. After one year of Tafamidis therapy, participants will return to initial facility where testing was preformed to undergo a follow up cardiac magnetic resonance imaging study.

There is emerging evidence that there may be biomarkers yet identified for earlier detection of this disease. Henceforth, investigators propose to collect and store blood samples for all participants for future analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they meet the following criteria:

  * 18 and 90 years of age
  * Transthyretin amyloid cardiomyopathy (ATTRwt or ATTRm) confirmed by genetic testing and/or presence of transthyretin precursor protein confirmed on immunohistochemical analysis, and/or scintigraphy
  * History of heart failure (NYHA I, II, or III)
  * Agreeable to treatment with Tafamidis

Exclusion Criteria:

* Patients will be excluded if any one of the following criteria are not met:

  * Heart failure not due to transthyretin amyloid cardiomyopathy
  * New York Heart Association (NYHA) class IV heart failure
  * Presence of light-chain amyloidosis (serum or urine)
  * Implanted cardiac device at baseline
  * Treatment with ATTR stabilizer or gene silencer within the past 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 131 patients diagnosed with ATTR-CM being treated with Tafamidis
Sampling Method: Non-Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Stabilization of Transthyretin Amyloid Cardiomyopathy | 1 year
  Stabilization as defined by reduction in extracellular volume on cardiac magnetic resonance after one year of Tafamidis therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No